CLINICAL TRIAL: NCT06701097
Title: The Effect of Emotion Regulation Training on the Levels of Alexithymia in Nursing College Students
Brief Title: Emotion Regulation Training, Nursing Student, and Alexithymia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Günay Öge, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E.60365
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Alexithymia; Emotion Regulation
Keywords: Alexithymia; Nursing; Emotion regulation; Student
MeSH Terms: conditions — Affective Symptoms; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emotion regulation training group (Experimental): Since the number of participants in the intervention group would prevent the training from being given as a group, the participants were divided into three different groups. Each group was given theoretical training on emotions, thoughts, physical symptoms resulting from emotions, and verbal and non-verbal ways of communicating emotions. The theoretical training was reinforced with activities such as relaxation exercises, role plays, imagination, brainstorming, etc. Each training lasted 60-90 minutes.
  Interventions: Behavioral: Emotion regulation training
- Control group (No Intervention): Participants in the control group did not receive any training. Only pre-test, post-test, and follow-up tests were applied to the individuals in this group.

INTERVENTIONS:
Behavioral: Emotion regulation training — Man is a social being and therefore interacts with his environment. In the process of interaction, they can transfer their feelings, thoughts, and information. However, the interaction process may not always continue smoothly. People's inability to express their emotions appropriately today negatively affects communication. The reason why people cannot express their emotions may be the high level of alexithymia. The concept of alexithymia means having difficulty in recognizing, expressing, and naming emotions. High levels of alexithymia in students, who are future healthcare professionals, can negatively affect themselves, other healthcare professionals and the patients they care for; it can cause burnout in healthcare professionals, decrease the quality of care they provide and cause them to experience interpersonal communication conflicts.
  Arms: Emotion regulation training group

SUMMARY:
This study aimed to investigate the effects of emotional regulation training, which is a prepared based on the cognitive behavioral approach, on alexithymia in nursing students.

DETAILED DESCRIPTION:
This study aimed to reduce alexithymia levels in nursing students with emotion regulation training based on a cognitive behavioral approach. The study was conducted with 74 nursing students, 37 in the intervention group and 37 in the control group, studying at a foundation university in the 2023-2024 academic year. The study data were collected using the data collection form and the Toronto Alexithymia Scale-20 (TAS-20). Data collection tools were applied three times as pre-post and follow-up tests. Male and female students who met the inclusion criteria of the study were determined by using the pre-test of the population. For the sample group to represent the population, students with high levels of alexithymia were identified by stratification by determining the class and gender ratios. Then, students were assigned to intervention and control groups by randomization. The 7-session training program prepared for the students in the intervention group was applied. No intervention was made to the control group during the implementation. After the training sessions were completed, post-test data were collected. Follow-up measurements were made three months later.

ELIGIBILITY:
Inclusion Criteria:

* To be a student of the nursing department
* Agree to participate in the study

Exclusion Criteria:

* Having received psychological support within the last 10 years
* Having a psychiatric disorder
* Not being a citizen of the Republic of Turkey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Toronto Alexithymia-20 Scale | - Before training. -immediately after the training is over. -Three months after training.
  The scale measures the alexithymia level of the individual. The scale is a Likert-type scale consisting of 20 items and scored between 1-5. The minimum score that can be obtained from the scale is 20 and the maximum score is 100. The higher the score obtained from the scale, the higher the alexithymia level of the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)